CLINICAL TRIAL: NCT03567759
Title: Effect 0ne Lung Ventilation and Open Pneumothorax on Respiratory Mechanics and Transpulmonary Pressure
Brief Title: Transpulmonary Pressure in One Lung Ventilation and Open Pneumothorax
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Amit Lehavi MD FANZCA, Director of Pediatric Anesthesia, Rambam Health Care Campus
Other Study IDs: RMB 15-0262
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Esophageal Pressure During one lung ventilation

DETAILED DESCRIPTION:
Esophageal pressure comparison during positive pressure ventilation, one lung ventilation, lateral position and open pneumothorax

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for VATS requiring one lung ventilation
* Body mass index below 35 kg/m^2

Exclusion Criteria:

* esophageal pathology preventing insertion of orogatric tube
* scoliosys

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients of age 18-85 years scheduled for VATS requiring one lung ventilation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in esophageal pressure | from tracheal intubation untill fiveminutes after induction of open pneumothorax
  esophageal pressure in supine and lateral positions, and following one lung ventilation and open pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Amit Lehavi, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel